CLINICAL TRIAL: NCT03920332
Title: Obstetric Outcomes of Women Suffering From Hereditary Fibrinogen Disorders
Brief Title: Pregnancy and Fibrinogen Disorders
Acronym: FIBRINOGEST
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Collaborators: Swiss Hemophilia Network (Other)
Responsible Party: Principal Investigator, Casini Alessandro, MD, Principal Investigator, University Hospital, Geneva
Other Study IDs: CCER2019-00353
Record Dates: First submitted 2019-04-12; First posted 2019-04-18 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Hypofibrinogenemia, Congenital; Afibrinogenemia, Congenital; Dysfibrinogenemia, Congenital
Keywords: Pregnancy; obstetric; miscarriage; haemorrhage; fibrinogen
MeSH Terms: conditions — Afibrinogenemia; Dysfibrinogenemia, Congenital; Abortion, Spontaneous; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this observational study is to evaluate the prevalence of uncomplicated pregnancies in women suffering from congenital fibrinogen disorders (i.e, hypofibrinogenemia, dysfibrinogenemia, hypodysfibrinogenemia) as well as to describe pregnancies outcomes in such diseases.

DETAILED DESCRIPTION:
Women with quantitative or qualitative fibrinogen disorders are often more prone to obstetrical complications, from bleeding to recurrent miscarriages or thrombosis. Data on fibrinogen levels variations throughout the pregnancy and on the delivery management are lacking. In this observational study will be include adult women with pas obstetrical history. A general questionnaire on demographics and clinical data will be filled out by the patient's physician. A detailed questionnaire on obstetrical data will also be completed contacting the patient in case of lacking data.

ELIGIBILITY:
Inclusion Criteria:

* Inherited fibrinogen disorders (hypofibrinogenemia, dysfibrinogenemia, hypodysfibrinogenemia)
* At lest one past pregnancy
* Adult

Exclusion Criteria:

* No past pregnancy
* Not confirmed fibrinogen disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women will be recruited in Hemophilia Centers.
Sampling Method: Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of normal issue pregnancy | At inclusion
  All pregnancy not resulting in miscarriage, stillbirth or abortion

SECONDARY OUTCOMES:
Prevalence of pregnancy without complications | At inclusion
  All pregnancy not resulting in intrauterine growth retardation, preterm labor, pregnancy-induced hypertension, gestational diabetes, preeclampsia, abruption placenta, anamniota, vaginal bleeding requiring medical intervention
Modalities of delivery | At inclusion
  Vaginal versus caesarean cut
Modalities of delivery | At inclusion
  Instrumental delivery vs none
Post-partum complications | At inclusion
  Post-partum haemorrhage and/or thrombotic event within 3 months after the delivery
Fibrinogen variations | At inclusion
  Fibrinogen levels throughout the pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Casini, MD, Principal Investigator — University Hospitals of Geneva; Justine Hugon-Rodin, MD, PHD, Principal Investigator — APHP
Locations (3):
- Hopital Port-Royal, Paris, France
- Jessenius Faculty of Medicine and University Hospital, Martin, Slovakia
- University Hospitals of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No